CLINICAL TRIAL: NCT00002477
Title: Phase III Randomized Study of Adjuvant Therapy With a Platinum-Containing Regimen (e.g., CBDCA or CAP: CTX/DOX/CDDP) vs No Adjuvant Therapy in Patients With Fully Resected Early Stage Ovarian Cancer
Brief Title: Adjuvant Chemotherapy Compared With Observation in Treating Patients With Resected Early Stage Ovarian Epithelial Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000077026; MRC-ICON1; EU-91002
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-07

CONDITIONS: Ovarian Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Doxorubicin

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of adjuvant therapy using platinum-based chemotherapy drugs with no adjuvant therapy in treating patients with early stage invasive ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether adjuvant chemotherapy with a platinum-containing regimen (e.g., carboplatin or CAP: cyclophosphamide/doxorubicin/cisplatin) prolongs survival in patients with early stage ovarian cancer compared to those receiving no adjuvant treatment.

OUTLINE: Randomized study. Patients are randomized to Arm I or II; treatment should begin within 6 weeks of surgery. Regimens listed in Arm I are recommended, but other platinum-containing regimens are allowed provided the doses at a minimum meet those listed below. Arm I: Single-agent Chemotherapy or 3-Drug Combination Chemotherapy. Carboplatin, CBDCA, NSC-241240; or CAP: Cyclophosphamide, CTX, NSC-26271; Doxorubicin, DOX, NSC-123127; Cisplatin, CDDP, NSC-119875. Arm II: Observation. No adjuvant therapy.

PROJECTED ACCRUAL: A maximum of 2,000 patients will be randomized.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed invasive ovarian cancer of epithelial origin All tumor resected prior to randomization Uncertain whether immediate chemotherapy is required

PATIENT CHARACTERISTICS: Age: Any age Performance status: Sufficient to receive chemotherapy Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No prior malignancy except nonmelanomatous skin cancer No clear contraindication to chemotherapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Minimum recommended surgical procedures (when possible): Thorough surgical staging Total hysterectomy/bilateral salpingo-oophorectomy Omentectomy, as follows: Total supracolonic omentectomy if omentum involved Removal of distal 2 cm or infracolonic omentectomy in the absence of macroscopic disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-04

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. Williams, DM, FRCP, Study Chair — Cochrane Cancer Network
Locations (1):
- Cochrane Cancer Network, Oxford, England, United Kingdom

REFERENCES:
- [Background] Colombo N, Trimbos JB, Guthrie D, et al.: ACTION + ICON1: two parallel randomised phase III trials comparing adjuvant chemotherapy to no adjuvant chemotherapy following surgery in women with high risk early ovarian cancer. [Abstract] Eur J Cancer 37 (suppl 6): A-1019, s276, 2001.
- [Result] Swart AC: Long-term follow-up of women enrolled in a randomized trial of adjuvant chemotherapy for early stage ovarian cancer (ICON1). [Abstract] J Clin Oncol 25 (Suppl 18): A-5509, 276s, 2007.
- [Result] Guthrie D: ICON1: a randomised trial of immediate platinum-based chemotherapy against chemotherapy delayed until indicated in women with ovarian cancer. [Abstract] Br J Cancer 85 (suppl 1): A-9.1, 28, 2001.
- [Result] Vergote IB, Trimbos BJ, Guthrie D, et al.: Results of a randomized trial in 923 patients with high-risk early ovarian cancer, comparing adjuvant chemotherapy with no further treatment following surgery. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-802, 2001.